CLINICAL TRIAL: NCT02572804
Title: A Randomised Controlled Trial of Thoracic Epidural Analgesia Versus Surgically Placed Rectus Sheath Catheters for Open Radical Cystectomy: Is There a Difference in Patient Outcomes?
Brief Title: Comparing Rectus Sheath Catheter to Epidural Post Cystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver Coastal Health (Other Government)
Collaborators: University of British Columbia (Other); Vancouver Prostate Centre (Other)
Responsible Party: Principal Investigator, Dr. Alan I. So, Urologic Surgeon, Vancouver Coastal Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V15-02041; H1502041 (Other: UBC CREB Number)
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Bladder Cancer; Postoperative Pain
Keywords: bladder cancer-cystectomy; rectus sheath catheter; epidural
MeSH Terms: conditions — Urinary Bladder Neoplasms; Pain, Postoperative | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectus Sheath Catheter Group (Active Comparator): Patients will have rectus sheath catheters surgically inserted with infusion of 0.125% Bupivicaine at 5mls an hour.
  Interventions: Device: Rectus Sheath Catheters
- Epidural Group (Active Comparator): Patients will have a standard epidural placement with infusion of 0.125% Bupivicaine at an initial rate of 5mls/hour, titrated to response
  Interventions: Device: Epidural

INTERVENTIONS:
Device: Epidural — Patients in this group will have an epidural inserted in a standard fashion, prior to the induction of anesthesia. These will be infused with 0.125% Bupivicaine at an initial rate of 5mls/hour, titrated to response. Patients will also receive a patient controlled analgesia with hydromorphone 0.2mg/ml, bolus of 200 micrograms with 6 minute lock out (variable in accordance with anesthetic preference).
  Arms: Epidural Group
Device: Rectus Sheath Catheters — Patients in this group will have surgically inserted rectus sheath catheters (bilaterally), immediately prior to closure of the anterior abdominal wall. These will be infused with 0.125% Bupivicaine at 5mls an hour at a standard rate.Patients will also receive a patient controlled analgesia with hydromorphone 0.2mg/ml, bolus of 200 micrograms with 6 minute lock out (variable in accordance with anesthetic preference).
  Arms: Rectus Sheath Catheter Group

SUMMARY:
This is a prospective randomised controlled trial that will compare the outcomes of rectus sheath catheters to epidurals in patients who have undergone a cystectomy, via a lower midline abdominal incision for bladder cancer.

DETAILED DESCRIPTION:
This study will compare the outcomes of two different pain control techniques, used as standard of care, following major abdominal surgery for bladder removal. Rectus sheath catheters are small tubes that are positioned into a specific area of the cut abdominal wall at the end of surgery; whereas an epidural is a tube that is positioned into the back. Both allow administration of local anaesthetic for pain control. The current gold standard is an epidural. This study will aim to evaluate this and show the comparative efficacy of the rectus sheath catheter, which anecdotally the investigators have found superior in practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients over or equal to the age of 19 years old who can understand the study protocol and are able to give consent
* Patients with an American Society of Anaesthesiology (ASA) classification 1 to 3
* Patients must have a preoperative oral 24 hour opioid consumption of less than or equal to 30mg morphine equivalents
* Patients must be able to understand and be able to use patient controlled analgesia
* Patients must be undergoing a cystectomy with an infra-umbilical midline incision

Exclusion Criteria:

* Patients with BMI greater than 40
* Patients with an allergy to local anaesthetics
* Patients who are contraindicated to having an epidural (e.g. coagulopathic, distorted anatomy, patient refusal, infection at the site of proposed insertion)
* Patients with previous spinal surgery at the proposed site of epidural
* Patients with neurodegenerative disorders or spinal cord injury
* Patients with known anatomy that would not permit placement of the rectus sheath catheters e.g. Prune Belly Syndrome
* Patients undergoing another complex abdominal procedure in addition to cystectomy and reconstruction requiring extension of the abdominal incision above the umbilicus.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative post-operative opioid consumption | To Day 3 post-op

SECONDARY OUTCOMES:
Visual Analogue Score pain score | within 4 hours post-operatively and on days 1, 2 and 3 post-operatively
Patient total intraoperative Opioid requirement | Intraoperatively
  Opioid requirement will be measured in morphine equivalents and reported as such on a per patient basis and measured throughout the operation.
Total patient fluid requirements throughout hospital admission | From the start of the operation to day 3 post-operatively.
  Measurement of individual patient fluid balance will be performed up to and including day 3 post-operatively.
Recorded evidence of hypotension | Until Day 3 postoperatively
  Hypotension for the purposes of this study is defined as a systolic blood pressure of less than 95.
Duration of post-operative ileus | This will be measured during the patients' inpatient hospital stay - usually up to a maximum of 10 days.
  Ileus will be measured by a 3 separate variables - bowel sounds, passing of flatus and opening of bowels. The post-operative day on which each of these targets is achieved for each patient will be recorded.
Time to mobilisation | The day at which patient achieves mobilisation - usually at a maximum of 5 days post-operatively
Length of Hospital Stay | The day at which patient is discharged from hospital- usually on average 10 days post-operatively
Patient Satisfaction with pain control | Day 3 post operatively
  Patient satisfaction with pain control will be measured using a 9-point Likert scale on day 3 post-operatively.
Complications and side effects. | 30 day morbidity and mortality
  At 30 days an electronic note review will be performed to evaluate for 30 day mortality and morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Martin E Gleave, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Prostate Centre, Dept. Urologic Sciences, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Bochner BH, Dalbagni G, Sjoberg DD, Silberstein J, Keren Paz GE, Donat SM, Coleman JA, Mathew S, Vickers A, Schnorr GC, Feuerstein MA, Rapkin B, Parra RO, Herr HW, Laudone VP. Comparing Open Radical Cystectomy and Robot-assisted Laparoscopic Radical Cystectomy: A Randomized Clinical Trial. Eur Urol. 2015 Jun;67(6):1042-1050. doi: 10.1016/j.eururo.2014.11.043. Epub 2014 Dec 8. PMID 25496767
- [Background] Block BM, Liu SS, Rowlingson AJ, Cowan AR, Cowan JA Jr, Wu CL. Efficacy of postoperative epidural analgesia: a meta-analysis. JAMA. 2003 Nov 12;290(18):2455-63. doi: 10.1001/jama.290.18.2455. PMID 14612482
- [Background] Rigg JR, Jamrozik K, Myles PS, Silbert BS, Peyton PJ, Parsons RW, Collins KS; MASTER Anaethesia Trial Study Group. Epidural anaesthesia and analgesia and outcome of major surgery: a randomised trial. Lancet. 2002 Apr 13;359(9314):1276-82. doi: 10.1016/S0140-6736(02)08266-1. PMID 11965272
- [Background] Ready LB. Acute pain: lessons learned from 25,000 patients. Reg Anesth Pain Med. 1999 Nov-Dec;24(6):499-505. doi: 10.1016/s1098-7339(99)90038-x. No abstract available. PMID 10588551
- [Background] Gustafsson UO, Hausel J, Thorell A, Ljungqvist O, Soop M, Nygren J; Enhanced Recovery After Surgery Study Group. Adherence to the enhanced recovery after surgery protocol and outcomes after colorectal cancer surgery. Arch Surg. 2011 May;146(5):571-7. doi: 10.1001/archsurg.2010.309. Epub 2011 Jan 17. PMID 21242424
- [Background] Guillotreau J, Game X, Mouzin M, Doumerc N, Mallet R, Sallusto F, Malavaud B, Rischmann P. Radical cystectomy for bladder cancer: morbidity of laparoscopic versus open surgery. J Urol. 2009 Feb;181(2):554-9; discussion 559. doi: 10.1016/j.juro.2008.10.011. Epub 2008 Dec 13. PMID 19084856
- [Background] Dutton TJ, McGrath JS, Daugherty MO. Use of rectus sheath catheters for pain relief in patients undergoing major pelvic urological surgery. BJU Int. 2014 Feb;113(2):246-53. doi: 10.1111/bju.12316. Epub 2013 Aug 13. PMID 23937574